CLINICAL TRIAL: NCT01544348
Title: A Phase 1 Randomized, Placebo-controlled, Dose-escalation Study to Evaluate the Safety of MEDI4212 in Subjects With IgE >= 30 IU/mL
Brief Title: A Phase 1, Randomized, Placebo-controlled, Dose-escalation Safety Study of MEDI4212 in Subjects With IgE >= 30 IU/mL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-RI-MEDI4212-1085
Record Dates: First submitted 2012-01-31; First posted 2012-03-05 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Allergic Asthma; Atopic Dermatitis; Allergic Rhinitis; Healthy Volunteers
Keywords: Allergic; Atopic Dermatitis; MEDI4212
MeSH Terms: conditions — Dermatitis, Atopic; Rhinitis, Allergic | interventions — Omalizumab; MEDI4212; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Placebo (Placebo Comparator): A single dose of placebo matched to MEDI4212 subcutaneous injection or intravenous infusion on Day 1.
  Interventions: Other: Placebo
- Omalizumab (Active Comparator): A single flexible dose of omalizumab between 150 to 375 milligram (mg) injection based upon participant's Immunoglobulin E (IgE) levels and body weight subcutaneously on Day 1.
  Interventions: Biological: Omalizumab
- MEDI4212 5 mg Subcutaneous (Experimental): A single dose of MEDI4212 5 mg injection subcutaneously on Day 1.
  Interventions: Biological: MEDI4212 5 mg Subcutaneous
- MEDI4212 15 mg Subcutaneous (Experimental): A single dose of MEDI4212 15 mg injection subcutaneously on Day 1.
  Interventions: Biological: MEDI4212 15 mg Subcutaneous
- MEDI4212 60 mg Subcutaneous (Experimental): A single dose of MEDI4212 60 mg injection subcutaneously on Day 1.
  Interventions: Biological: MEDI4212 60 mg Subcutaneous
- MEDI4212 150 mg Subcutaneous (Experimental): A single dose of MEDI4212 150 mg injection subcutaneously on Day 1.
  Interventions: Biological: MEDI4212 150 mg Subcutaneous
- MEDI4212 300 mg Subcutaneous (Experimental): A single dose of MEDI4212 300 mg injection subcutaneously on Day 1.
  Interventions: Biological: MEDI4212 300 mg Subcutaneous
- MEDI4212 300 mg Intravenous (Experimental): A single dose of MEDI4212 300 mg intravenous infusion over 120 minutes on Day 1.
  Interventions: Biological: MEDI4212 300 mg Intravenous

INTERVENTIONS:
Other: Placebo — A single dose of placebo matched to MEDI4212 subcutaneous injection or intravenous infusion on Day 1.
  Arms: Placebo
Biological: Omalizumab — A single flexible dose of omalizumab between 150 to 375 milligram (mg) injection based upon participant's Immunoglobulin E (IgE) levels and body weight subcutaneously on Day 1.
  Other Names: Xolair
  Arms: Omalizumab
Biological: MEDI4212 5 mg Subcutaneous — A single dose of MEDI4212 5 mg injection subcutaneously on Day 1.
  Arms: MEDI4212 5 mg Subcutaneous
Biological: MEDI4212 15 mg Subcutaneous — A single dose of MEDI4212 15 mg injection subcutaneously on Day 1.
  Arms: MEDI4212 15 mg Subcutaneous
Biological: MEDI4212 60 mg Subcutaneous — A single dose of MEDI4212 60 mg injection subcutaneously on Day 1.
  Arms: MEDI4212 60 mg Subcutaneous
Biological: MEDI4212 150 mg Subcutaneous — A single dose of MEDI4212 150 mg injection subcutaneously on Day 1.
  Arms: MEDI4212 150 mg Subcutaneous
Biological: MEDI4212 300 mg Subcutaneous — A single dose of MEDI4212 300 mg injection subcutaneously on Day 1.
  Arms: MEDI4212 300 mg Subcutaneous
Biological: MEDI4212 300 mg Intravenous — A single dose of MEDI4212 300 mg intravenous infusion over 120 minutes on Day 1.
  Arms: MEDI4212 300 mg Intravenous

SUMMARY:
Phase 1 study to evaluate the safety of MEDI4212.

DETAILED DESCRIPTION:
A Phase 1, randomized, placebo-controlled, dose-escalation study to evaluate the safety and tolerability of ascending single subcutaneous and intravenous doses of MEDI4212 in subjects with immunoglobulin E (IgE) greater than or equal to (>=) 30 international units per milliliters (IU/mL).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 60 years
* Written informed consent and any locally required authorization
* Body weight 45-150 kilogram (kg) for Cohorts 1-3, 4b, and 5-9. Body weight 45-90 kg for Cohort 4a
* Females must have been surgically sterilized or postmenopausal
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from Day 1 through Day 85; Both partners to use contraception
* Sterilized males must be at least 1-year post vasectomy or use a highly effective contraceptive method
* Healthy Japanese population as determined by a responsible physician
* Current diagnosis of allergic rhinitis, allergic asthma, or atopic dermatitis (cohorts 1-6) with a diagnostic immunoglobulin E (IgE) of 30 international units per milliliter (IU/mL) at Screening. Diagnostic IgE levels are further restricted for subjects enrolling into each cohort, with the following levels required at Screening: Cohorts 1 and 2: 30-700 IU/mL; Cohort 3: 30-700 IU/mL (4 subjects), greater than (>) 700-1,200 IU/mL (4 subjects), and >1,200 IU/mL (4 subjects); Cohort 4a: 30-500 IU/mL; Cohort 4b: >700 IU/mL; Cohorts 5 and 6: 30-700 IU/mL (4 subjects per cohort) and >700 IU/mL (6 subjects per cohort) or Japanese Cohorts 7-9: greater than or equal to (>=) 30 IU/mL
* Nonsmoker for >=6 months
* Obsolete criteria as no longer require Positive in vitro IgE fluorescence enzyme immunoassay (FEIA) response
* A forced expiration volume in one second (FEV1) >= 80 percent (%) predicted in subjects with asthma. Non-asthmatic subjects with FEV1 >=80% predicted, or with FEV1 less than (<) 80% predicted but who, in the opinion of the investigator, do not have lung disease
* Ability and willingness to complete the follow-up period through Day 85 as required by the protocol.

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Concurrent enrollment in another clinical study
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals
* Exposure to an anti-IgE monoclonal antibodies (MAb) within 12 months prior to Screening
* Positive drug screen at Screening or Day -1. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines
* History of regular alcohol abuse within 12 months prior to Screening
* History of sensitivity to any component of the investigational product formulation or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation
* Subjects with abnormal liver function test values (aspartate transaminase [AST] and alanine transaminase [ALT]) at Screening as defined as follows: a) Liver function test values >= 1.5 times upper limit of normal (ULN)
* Unwillingness or inability to follow the procedures outlined in the protocol
* Positive test or history of hepatitis B or positive hepatitis C
* Positive test or history of human immunodeficiency virus (HIV) or subject is known to be HIV seropositive
* History of cancer, with the exception of basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success
* Women who are pregnant, breastfeeding, or lactating
* Plans to donate blood during the study period
* Hyper-IgE syndrome or bronchopulmonary aspergillosis
* Prior history of Immune Complex Disease or type 3 hypersensitivity reactions to MAb administration
* Known history of prior infusion reaction to MAb administration
* History of untreated parasitic/helminthic infection within 6 months prior to Screening
* Uses any of the following medications: a) Oral corticosteroids b) Medium to high dose Immunocorticosteroids (ICS)/ long-acting beta agonists (LABA) c) Immunosuppressives d) Beta blockers
* If receiving allergy immunotherapy, must be on stable dose for 3 months. Must not receive allergy immunotherapy within 7 days of investigational product administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 295 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site, Cypress, California
  - Research Site, Glendale, California
  - Research Site, Denver, Colorado
  - Research Site, Miami, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Madison, Wisconsin

REFERENCES:
- [Derived] Sheldon E, Schwickart M, Li J, Kim K, Crouch S, Parveen S, Kell C, Birrell C. Pharmacokinetics, Pharmacodynamics, and Safety of MEDI4212, an Anti-IgE Monoclonal Antibody, in Subjects with Atopy: A Phase I Study. Adv Ther. 2016 Feb;33(2):225-51. doi: 10.1007/s12325-016-0287-8. Epub 2016 Feb 3. PMID 26843086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 295 participants were screened, out of which 209 were screen failures and 86 were randomized.
Period: Overall Study
Arm/Group | Placebo | Omalizumab | MEDI4212 5 mg Subcutaneous | MEDI4212 15 mg Subcutaneous | MEDI4212 60 mg Subcutaneous | MEDI4212 150 mg Subcutaneous | MEDI4212 300 mg Subcutaneous | MEDI4212 300 mg Intravenous
Started | 17 | 6 | 3 | 3 | 16 | 19 | 14 | 8
Treated | 17 | 6 | 3 | 3 | 15 | 18 | 14 | 8
Completed | 15 | 6 | 3 | 3 | 15 | 16 | 12 | 8
Not Completed | 2 | 0 | 0 | 0 | 1 | 3 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of investigational product and had safety data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab | MEDI4212 5 mg Subcutaneous | MEDI4212 15 mg Subcutaneous | MEDI4212 60 mg Subcutaneous | MEDI4212 150 mg Subcutaneous | MEDI4212 300 mg Subcutaneous | MEDI4212 300 mg Intravenous | Total
Number analyzed (Participants) | 17 | 6 | 3 | 3 | 15 | 18 | 14 | 8 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (12.6) | 39.3 (9.2) | 44.7 (3.2) | 40.3 (9.6) | 38.7 (12.5) | 40.3 (11.1) | 35.9 (13.1) | 38.0 (8.6) | 39.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 1 | 2 | 4 | 4 | 2 | 0 | 22
  Male | 10 | 4 | 2 | 1 | 11 | 14 | 12 | 8 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study drug and up to Day 85 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 to 85
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab | MEDI4212 5 mg Subcutaneous | MEDI4212 15 mg Subcutaneous | MEDI4212 60 mg Subcutaneous | MEDI4212 150 mg Subcutaneous | MEDI4212 300 mg Subcutaneous | MEDI4212 300 mg Intravenous
Number analyzed (Participants) | 17 | 6 | 3 | 3 | 15 | 18 | 14 | 8
participants
  TEAEs | 8 | 2 | 2 | 1 | 4 | 9 | 7 | 6
  TESAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Observed Serum Concentration
Description: Serum concentration of omalizumab and MEDI4212 were measured for participants who received omalizumab and MEDI4212, respectively.
Time Frame: Pre-dose and post-dose on Day 1; Day 2, 3, 5, 8, 15, 22, 29, 43, 57 and 85
Population: Pharmacokinetic (PK) population included all participants who received any investigational product and had a sufficient number of serum concentration measurements for computing PK parameters. Here 'n' signifies participants evaluable for this outcome measure at specified time point, for each group respectively
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Omalizumab | MEDI4212 5 mg Subcutaneous | MEDI4212 15 mg Subcutaneous | MEDI4212 60 mg Subcutaneous | MEDI4212 150 mg Subcutaneous | MEDI4212 300 mg Subcutaneous | MEDI4212 300 mg Intravenous
Number analyzed (Participants) | 6 | 3 | 3 | 15 | 18 | 14 | 8
nanogram per milliliter (ng/mL)
  Day 1 (predose) (n=0,1,0,0,2,1,1) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 96.76 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 254.71 (134.58) | 91.69 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 158.32 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  Day 1 (postdose) (n=0,0,0,0,0,0,8) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 110693 (26060.2)
  Day 2 (n=5,1,1,12,17,13,8) | 8941.12 (6361.95) | 100.36 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 292.76 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 3146.54 (3820.61) | 6108.21 (3401.45) | 14971.9 (9608.63) | 88457.0 (23398.4)
  Day 3 (n=5,1,1,12,17,14,8) | 13912.4 (7546.50) | 110.12 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 312.73 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 3131.79 (2513.43) | 7969.07 (4004.75) | 14771 (8692.16) | 69776.5 (37738.7)
  Day 5 (n=5,1,1,11,16,14,8) | 17016.3 (6806.15) | 116.44 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 284.28 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 3336.31 (2759.69) | 7227.93 (3210.9) | 15183.4 (8522.98) | 34359.5 (6817.40)
  Day 8 (n=5,0,1,9,16,14,8) | 16467.4 (5374.97) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 190.38 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 2368.21 (1364.28) | 7144.03 (5078.61) | 12611.1 (8382.56) | 39290.2 (32657.3)
  Day 15 (n=5,0,0,7,14,13,8) | 15099.6 (5470.44) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 1134.39 (259.41) | 4514.83 (2864.46) | 8824.94 (6744.55) | 11391.2 (3673.21)
  Day 22 (n=5,0,0,6,12,10,8) | 12780.2 (4657.23) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 521.3 (96.73) | 3401 (2140.78) | 7454.01 (4682.86) | 4644.04 (2571.96)
  Day 29 (n=5,0,0,4,11,8,7) | 9466.26 (4040.07) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 212.22 (82.96) | 2176.59 (1390.94) | 2688.85 (2191.8) | 2045.55 (1814.12)
  Day 43 (n=5,2,0,0,5,5,3) | 5195.21 (2263.08) | 121.39 (8.11) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 1544.4 (2068.43) | 1188.63 (949.33) | 1669.74 (739.22)
  Day 57 (n=5,2,0,0,4,4,3) | 2367.85 (984.70) | 122.00 (0.35) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 290.44 (228.81) | 485.18 (249.73) | 150.90 (87.96)
  Day 85 (n=5,2,0,1, 3,1,1) | 829.55 (434.33) | 104.07 (2.48) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 98.62 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 202.54 (107.75) | 84.03 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 176.87 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

3. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies for MEDI4212 at Any Visit
Description: Anti-drug antibodies for MEDI4212 were analyzed for participants who received placebo or MEDI4212 as per planned analysis.
Time Frame: Days 1 (pre-dose), 15, 43, and 85
Population: Immunogenicity population included all participants who received any investigational product and had at least one valid immunogenicity test result.
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI4212 5 mg Subcutaneous | MEDI4212 15 mg Subcutaneous | MEDI4212 60 mg Subcutaneous | MEDI4212 150 mg Subcutaneous | MEDI4212 300 mg Subcutaneous | MEDI4212 300 mg Intravenous
Number analyzed (Participants) | 17 | 3 | 3 | 15 | 18 | 14 | 8
participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Free Immunoglobulin E (IgE) Serum Concentration
Time Frame: Day -28 (Screening), -1, 1 (pre-dose), 2, 3, 5, 8, 15, 22, 29, 43, 57, and 85 for all groups; 2 hours post-dose on Day 1 for MEDI4212 300 mg Intravenous group only
Population: Safety population included all participants who received any amount of investigational product and had safety data available. 'n' signifies those participants who evaluable for this outcome measure at specified time point for each group, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Omalizumab | MEDI4212 5 mg Subcutaneous | MEDI4212 15 mg Subcutaneous | MEDI4212 60 mg Subcutaneous | MEDI4212 150 mg Subcutaneous | MEDI4212 300 mg Subcutaneous | MEDI4212 300 mg Intravenous
Number analyzed (Participants) | 17 | 6 | 3 | 3 | 15 | 18 | 14 | 8
ng/mL
  Day -28 (n=16,6,3,3,14,15,13,8) | 1160.79 (1402.74) | 478.99 (369.31) | 655.76 (240.78) | 601.40 (342.13) | 2170.63 (3899.67) | 1976.98 (3172.11) | 1775.68 (2558.08) | 2641.68 (2332.13)
  Day -1 (n=17,6,3,3,15,17,14,7) | 1025.19 (1287.86) | 296.73 (185.09) | 589.62 (175.14) | 522.23 (259.96) | 2453.85 (3795.64) | 1655.06 (2866.87) | 1681.82 (2161.25) | 2772.55 (2320.93)
  Day 1 (Predose) (n=17,6,3,3,15,17,14,8) | 1155.59 (1447.09) | 410.78 (289.39) | 552.30 (168.96) | 558.69 (305.68) | 2754.09 (4468.96) | 1910.45 (3268.58) | 1850.27 (2435.13) | 2426.66 (2460.85)
  Day 1:2 hours postdose (n=0,0,0,0,0,0,0,8) | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | NA (NA) — No participant was evaluable for this outcome measure at this time point. | 0.00 (0.00)
  Day 2 (n=17,6,3,3,15,17,14,8) | 1183.10 (1494.92) | 71.89 (157.68) | 302.31 (195.18) | 336.75 (294.36) | 1584.76 (3999.13) | 366.83 (1499.49) | 94.19 (351.27) | 0.00 (0.00)
  Day 3 (n=17,6,3,3,15,17,14,8) | 1175.50 (1550.93) | 74.29 (168.46) | 282.12 (179.53) | 293.78 (259.88) | 1366.58 (3496.19) | 248.20 (1022.97) | 42.24 (157.38) | 0.00 (0.00)
  Day 5 (n=17,6,3,3,15,17,14,8) | 1131.87 (1448.24) | 74.85 (169.36) | 297.90 (193.62) | 277.94 (240.84) | 1401.33 (3429.60) | 253.71 (1045.75) | 0.53 (1.43) | 0.00 (0.00)
  Day 8 (n=17,6,3,3,15,17,14,8) | 1119.38 (1417.95) | 85.00 (192.16) | 366.17 (239.65) | 288.20 (250.03) | 1704.44 (3822.59) | 362.27 (1408.50) | 3.17 (10.71) | 0.00 (0.00)
  Day 15 (n=17,6,3,3,15,17,14,8) | 1081.11 (1338.94) | 74.94 (161.38) | 418.27 (193.63) | 362.06 (246.96) | 2102.53 (4140.14) | 978.17 (2490.21) | 209.71 (539.11) | 0.00 (0.00)
  Day 22 (n=17,6,3,3,15,17,14,8) | 1084.02 (1294.17) | 70.95 (145.36) | 453.89 (191.07) | 406.12 (264.19) | 2111.36 (3730.60) | 1351.52 (2803.98) | 788.30 (1783.50) | 0.32 (0.60)
  Day 29 (n=16,6,3,3,15,17,13,8) | 1185.82 (1379.20) | 74.02 (143.04) | 478.53 (196.36) | 403.17 (232.44) | 2153.91 (3376.54) | 1676.12 (3296.43) | 1468.72 (3043.16) | 497.42 (628.41)
  Day 43 (n=16,6,3,3,15,16,13,8) | 1089.90 (1306.97) | 89.32 (157.95) | 496.28 (179.01) | 510.78 (301.83) | 2712.59 (4065.37) | 1928.37 (3371.88) | 1912.71 (2966.45) | 1674.54 (1689.61)
  Day 57 (n=16,6,3,3,15,15,12,8) | 1055.20 (1257.08) | 105.46 (159.88) | 506.63 (205.91) | 503.33 (326.80) | 2201.38 (3609.05) | 1394.92 (2394.88) | 2306.44 (3511.87) | 1978.31 (1906.57)
  Day 85 (n=15,6,3,3,15,16,12,8) | 913.17 (1142.25) | 294.89 (377.39) | 526.93 (227.80) | 530.49 (292.24) | 2014.95 (2952.69) | 1749.34 (2799.68) | 2528.85 (3967.57) | 2055.68 (1822.85)

ADVERSE EVENTS:
Time Frame: Day 1 to 85
Description: Safety population included all participants who received any amount of investigational product and had safety data available.
Arm/Group | Placebo | Omalizumab | MEDI4212 5 mg Subcutaneous | MEDI4212 15 mg Subcutaneous | MEDI4212 60 mg Subcutaneous | MEDI4212 150 mg Subcutaneous | MEDI4212 300 mg Subcutaneous | MEDI4212 300 mg Intravenous
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/6 | 0/3 | 0/3 | 0/15 | 0/18 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 8/17 | 2/6 | 2/3 | 1/3 | 4/15 | 9/18 | 7/14 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Omalizumab (N=6) | MEDI4212 5 mg Subcutaneous (N=3) | MEDI4212 15 mg Subcutaneous (N=3) | MEDI4212 60 mg Subcutaneous (N=15) | MEDI4212 150 mg Subcutaneous (N=18) | MEDI4212 300 mg Subcutaneous (N=14) | MEDI4212 300 mg Intravenous (N=8)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.